CLINICAL TRIAL: NCT04501679
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Nemolizumab (CD14152) in Subjects With Prurigo Nodularis
Brief Title: A Study to Assess the Efficacy and Safety of Nemolizumab (CD14152) in Participants With Prurigo Nodularis (PN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.203065; 2019-004789-17 (EudraCT Number)
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Prurigo Nodularis
Keywords: Prurigo; Neurodermatitis; Pruritus; Skin diseases
MeSH Terms: conditions — Prurigo; Neurodermatitis; Pruritus; Skin Diseases | interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nemolizumab (Experimental): Participants weighing less than (<) 90 kilogram (kg) received two subcutaneous (SC) injections of 30 milligrams (mg) nemolizumab (60 mg loading dose) at baseline then one SC injection once for every 4 weeks (Q4W). Participants weighing greater than or equal to (>=) 90 kg received two SC injections of 30 mg nemolizumab (60 mg total) at baseline (no loading dose) and two SC injections Q4W throughout the treatment period of 16 weeks.
  Interventions: Drug: Nemolizumab
- Placebo (Placebo Comparator): Participants weighing < 90 kg received two SC injections of matching placebo at baseline, then one SC injection Q4W. Participants weighing >= 90 kg received two SC injections of matching placebo at baseline, then two SC injections Q4W throughout the treatment period of 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nemolizumab — Participants received either 30 mg or 60 mg dose of nemolizumab as SC injection.
  Other Names: CD14152
  Arms: Nemolizumab
Drug: Placebo — Participants received matching placebo as SC injection.
  Arms: Placebo

SUMMARY:
The primary objective was to assess the efficacy of nemolizumab (CD14152) compared to placebo in participants greater than or equal to (>=) 18 years of age with prurigo nodularis (PN) after a 16-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PN for at least 6 months with: Pruriginous nodular lesions on upper limbs, trunk, and/or lower limbs, at least 20 nodules on the entire body with a bilateral distribution and Investigator Global Assessment (IGA) score more than equal to (>=) 3 (based on the IGA scale ranging from 0 to 4, in which 3 was moderate and 4 is severe) at both the screening and baseline visits
* Severe pruritus was defined as follows on the PP NRS:

  1. At the screening visit (Visit 1): PP NRS score was >= 7.0 for the 24-hour period immediately preceding the screening visit.
  2. At the baseline visit (Visit 2): Mean of the daily intensity of the PP NRS score was >= 7.0 over the previous week
* Female participants of childbearing potential (that is [i.e,], fertile, following menarche and until becoming post-menopausal unless permanently sterile) must agree to use at least 1 adequate and approved method of contraception throughout the study and for 12 weeks after the last study drug injection

Exclusion Criteria:

* Body weight less than < 30 kg
* Chronic pruritus resulting from another active condition other than PN, such as but not limited to scabies, lichen simplex chronicus, psoriasis, atopic dermatitis, contact dermatitis, acne, folliculitis, lichen planus, habitual picking/excoriation disorder, sporotrichosis, bullous autoimmune disease, end-stage renal disease, or cholestatic liver disease (example [eg] primary biliary cirrhosis) or diabetes mellitus or thyroid disease that is not adequately treated, as per standard of care
* Unilateral lesions of prurigo (eg, only one arm affected)
* History of or current confounding skin condition (eg, Netherton syndrome, cutaneous T-cell lymphoma [mycosis fungoides or Sezary syndrome], chronic actinic dermatitis, dermatitis herpetiformis)
* Participants with a current medical history of chronic obstructive pulmonary disease and/or chronic bronchitis
* Neuropathic and psychogenic pruritus such as but not limited to notalgia paresthetica, brachioradial pruritus, small fiber neuropathy, skin picking syndrome, or delusional parasitosis
* Requiring rescue therapy for PN during the screening period or expected to require rescue therapy within 4 weeks following the baseline visit
* Positive serology results (hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb], hepatitis C (HCV) antibody with positive confirmatory test for HCV (eg, polymerase chain reaction [PCR]), or human immunodeficiency virus antibody) at the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (22):
  - Galderma Investigational Site, Fountain Valley, California
  - Galderma Investigational Site, San Diego, California
  - Galderma Investigational Site, Washington D.C., District of Columbia
  - Galderma Investigational Site, Aventura, Florida
  - Galderma Investigational Site, Miami, Florida
  - Galderma Investigational Site, North Miami Beach, Florida
  - Galderma Investigational Site, Ormond Beach, Florida
  - Galderma Investigational Site, Chicago, Illinois
  - Galderma Investigational Site, Indianapolis, Indiana
  - Galderma Investigational Site, Louisville, Kentucky
  - Galderma Investigational Site, Boston, Massachusetts
  - Galderma Investigational Site, Saint Joseph, Michigan
  - Galderma Investigational Site, New York, New York
  - Galderma Investigational Site, Cincinnati, Ohio
  - Galderma Investigational Site, Dublin, Ohio
  - Galderma Investigational Site, Anderson, South Carolina
  - Galderma Investigational Site, Murfreesboro, Tennessee
  - Galderma Investigational Site, Dallas, Texas
  - Galderma Investigational Site, Dripping Springs, Texas
  - Galderma Investigational Site, Pflugerville, Texas
  - Galderma Investigational Site, Webster, Texas
  - Galderma Investigational Site, Morgantown, West Virginia
- Belgium (5):
  - Galderma Investigational Site, Brussels
  - Galderma Investigational Site, Ghent
  - Galderma Investigational Site, Jette
  - Galderma Investigational Site, Leuven
  - Galderma Investigational Site, Liège
- Canada (5):
  - Galderma Investigational Site, North York, Ontario
  - Galderma Investigational Site, Bathurst
  - Galderma Investigational Site, Calgary
  - Galderma Investigational Site, London
  - Galderma Investigational Site, Markham
- France (11):
  - Galderma Investigational Site, Bordeaux
  - Galderma Investigational Site, Brest
  - Galderma Investigational Site, Lille
  - Galderma Investigational Site, Nantes
  - Galderma Investigational Site, Nice
  - Galderma Investigational Site, Paris
  - Galderma Investigational Site, Pierre-Bénite
  - Galderma Investigational Site, Rouen
  - Galderma Investigational Site, Saint-Etienne
  - Galderma Investigational Site, Toulouse
  - Galderma Investigational Site, Valence
- Netherlands (2):
  - Galderma Investigational Site, Groningen
  - Galderma Investigational Site, Utrecht
- Poland (11):
  - Galderma Investigational Site, Bydgoszcz
  - Galderma Investigational Site, Chorzów
  - Galderma Investigational Site, Krakow
  - Galderma Investigational Site, Lodz
  - Galderma Investigational Site, Lublin
  - Galderma Investigational Site, Olsztyn
  - Galderma Investigational Site, Ostrowiec Świętokrzyski
  - Galderma Investigational Site, Rzeszów
  - Galderma Investigational Site, Szczecin
  - Galderma Investigational Site, Warsaw
  - Galderma Investigational Site, Wroclaw
- South Korea (2):
  - Galderma Investigational Site, Gyeonggi-do
  - Galderma Investigational Site, Seoul
- Spain (2):
  - Galderma Investigational Site, Barcelona
  - Galderma Investigational Site, Las Palmas de Gran Canaria
- Switzerland (5):
  - Galderma Investigational Site, Bern
  - Galderma Investigational Site, Buochs
  - Galderma Investigational Site, Lausanne
  - Galderma Investigational Site, Sankt Gallen
  - Galderma Investigational Site, Weinfelden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized data sets from which results presented are derived.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data availability will begin 6 months after approval of the indication by a regulatory body.
  Data availability will end 5 years from publication of the primary study results article.
Access Criteria: Data will be made available to qualified science and medical researchers upon formal request and submission of research proposal detailing planned analyses. Proposals should be directed to clinical.studies@galderma.com

REFERENCES:
- [Result] Kwatra SG, Yosipovitch G, Legat FJ, Reich A, Paul C, Simon D, Naldi L, Lynde C, De Bruin-Weller MS, Nahm WK, Sauder M, Gharib R, Barbarot S, Szepietowski JC, Conrad C, Fleischer A, Laquer VT, Misery L, Serra-Baldrich E, Lapeere H, Ahmad F, Jabbar Lopez ZK, Piketty C, Stander S; OLYMPIA 2 Investigators. Phase 3 Trial of Nemolizumab in Patients with Prurigo Nodularis. N Engl J Med. 2023 Oct 26;389(17):1579-1589. doi: 10.1056/NEJMoa2301333. PMID 37888917
- [Derived] Stander S, Rodriguez DN, Dias-Barbosa C, Filipenko D, Puelles J, Jabbar-Lopez ZK, Piketty C, Wiegmann H, Kwatra SG. Content Validity and Psychometric Validation of an Adapted Version of the Subject Sleep Diary in Prurigo Nodularis. Dermatol Ther (Heidelb). 2025 Jun;15(6):1405-1426. doi: 10.1007/s13555-025-01406-1. Epub 2025 Apr 23. PMID 40266487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 55 sites in 9 countries.
Pre-assignment Details: A total of 274 participants were randomized and treated (183 participants in Nemolizumab and 91 participants in Placebo group) received treatment in this study.
Period: Overall Study
Arm/Group | Nemolizumab | Placebo
Started | 183 | 91
Treated | 183 | 91
Completed | 174 | 88
Not Completed | 9 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Nemolizumab: Participants weighing <90 kg received two SC injections of 30 mg nemolizumab (60 mg loading dose) at baseline then one SC injection Q4W. Participants weighing >=90 kg received two SC injections of 30 mg nemolizumab (60 mg total) at baseline (no loading dose) and two SC injections Q4W throughout the treatment period of 16 weeks.
  Nemolizumab: Participants received either 30 mg or 60 mg dose of nemolizumab as SC injection.
- Placebo: Participants weighing <90 kg received two SC injections of matching placebo at baseline, then one SC injection Q4W. Participants weighing >=90 kg received two SC injections of matching placebo at baseline, then two SC injections Q4W throughout the treatment period of 16 weeks.
  Placebo: Participants received matching placebo as SC injection.
- Total: Total of all reporting groups
Arm/Group | Nemolizumab | Placebo | Total
Number analyzed (Participants) | 183 | 91 | 274
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (14.41) | 50.8 (15.00) | 52.7 (14.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 55 | 168
  Male | 70 | 36 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 173 | 79 | 252
  Unknown or Not Reported | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 23 | 14 | 37
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 5 | 7 | 12
  White | 147 | 68 | 215
  More than one race | 0 | 0 | 0
  Others | 5 | 2 | 7
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 122 | 61 | 183
  North America | 47 | 22 | 69
  Pacifica | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Improvement of Greater Than or Equal to (>=) 4 From Baseline in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 16
Description: The Peak Pruritus NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores were provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome. Weekly values are calculated as average of 7 consecutive days data up to the target study day (excluding) and set to missing, if less than 4 days data are available. Analysis window extension was applied to both timepoints, as described in the SAP. If a subject received any rescue therapy, the data at/after receipt of rescue therapy are considered as non-responders. Subjects with missing results are considered as non-responders.
Time Frame: Baseline, Week 16
Population: ITT population consisted of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 183 | 91
Participants | 103 | 19
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures were reported and continued when previous outcome measure was statistically significant at two-sided 0.05; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — A 2-sided p-value was derived from Cochran-Mantel-Haenszel (CMH) test using the randomized stratification variables (analysis center and body weight at randomization [< 90 kg, >= 90 kg]). Threshold of significance at 0.05; Cochran-Mantel-Haenszel (CMH) test using the randomized stratification variables (analysis center and body weight at randomization [<90 kg,>=90 kg]); Strata-adjusted percentage difference = 37.4, 95% CI 2-sided [26.3 to 48.5] — Strata adjusted percentage difference was obtained using weighted average of stratum-specific percentage using CMH

2. Primary Outcome: Number of Participants With an Investigator Global Assessment (IGA) Success at Week 16
Description: IGA success is defined as clear (0) or almost clear (1), and a reduction from baseline of greater than or equal to 2 points at week 16. Full scale is scored from 0-4, higher score indicates more severe symptoms. If a subject received any rescue therapy, the data at/after receipt of rescue therapy are considered as non-responders. Subjects with missing results are considered as non-responders.
Time Frame: Baseline, Week 16
Population: ITT population consisted of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 183 | 91
Participants | 69 | 10
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 28.5, 95% CI 2-sided [18.8 to 38.2] — Strata adjusted percentage difference was obtained using weighted average of stratum-specific percentage using CMH

3. Secondary Outcome: Number of Participants With an Improvement of >= 4 From Baseline in Weekly Average PP NRS at Week 4
Description: The Peak Pruritus NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores were provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome. Weekly values are calculated as average of 7 consecutive days data up to the target study day (excluding) and set to missing, if less than 4 days data are available. Analysis window extension was applied to baseline, as described in the SAP. If a subject received any rescue therapy, the data at/after receipt of rescue therapy are considered as non-responders. Subjects with missing results are considered as non-responders.
Time Frame: Baseline, Week 4
Population: ITT population consisted of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 183 | 91
Participants | 75 | 7
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 33.4, 95% CI 2-sided [24.3 to 42.4] — Strata adjusted percentage difference was obtained using weighted average of stratum-specific percentage using CMH

4. Secondary Outcome: Number of Participants With PP NRS < 2 at Week 16
Description: The Peak Pruritus NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores were provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome. Weekly values are calculated as average of 7 consecutive days data up to the target study day (excluding) and set to missing, if less than 4 days data are available. Analysis window extension was applied to week 16, as described in the SAP. If a subject received any rescue therapy, the data at/after receipt of rescue therapy are considered as non-responders. Subjects with missing results are considered as non-responders.
Time Frame: Week 16
Population: ITT population consisted all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 183 | 91
Participants | 64 | 7
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; CMH test using the randomized stratification variables (analysis center and body weight at randomization [<90 kg,>=90 kg]); Strata-adjusted percentage difference = 30.0, 95% CI 2-sided [21.3 to 38.6] — Strata adjusted percentage difference was obtained using weighted average of stratum-specific percentage using CMH

5. Secondary Outcome: Number of Participants With an Improvement of >=4 From Baseline in Sleep Disturbance Numeric Rating Scale (SD NRS) at Week 16
Description: The SD NRS is a scale to be used by the participants to report the degree of their sleep loss related to PN. The baseline SD NRS was determined based on the average of daily SD NRS (score ranging from 0 to 10) during the 7 days up to the treatment start (including until treatment start time) (rounding to nearest whole number is not permitted). A minimum of 4 daily scores out of the 7 days up to baseline study day is required for this calculation. On a scale of 0 to 10, with 0 being 'no sleep loss related to the symptoms of my skin disease (prurigo nodularis)' and 10 being 'I did not sleep at all due to the symptoms of prurigo nodularis'. Higher scores indicate worse outcome. Analysis window extension was applied to both timepoints, as described in the SAP. If a subject received any rescue therapy, the data at/after receipt of rescue therapy are considered as non-responders. Subjects with missing results are considered as non-responders.
Time Frame: Baseline, Week 16
Population: ITT population consisted all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 183 | 91
Participants | 95 | 19
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 4, analysis 1]; Strata-adjusted percentage difference = 31.9, 95% CI 2-sided [20.7 to 43.2] — Strata adjusted percentage difference was obtained using weighted average of stratum-specific percentage using CMH

6. Secondary Outcome: Number of Participants With an Improvement of >=4 From Baseline in SD NRS at Week 4
Description: The SD NRS is a scale to be used by the participants to report the degree of their sleep loss related to PN. The baseline SD NRS was determined based on the average of daily SD NRS (score ranging from 0 to10) during the 7 days up to the treatment start (including until treatment start time) (rounding to nearest whole number is not permitted). A minimum of 4 daily scores out of the 7 days up to baseline study day is required for this calculation. On a scale of 0 to 10, with 0 being 'no sleep loss related to the symptoms of my skin disease (prurigo nodularis)' and 10 being 'I did not sleep at all due to the symptoms of prurigo nodularis'. Higher scores indicate worse outcome. Analysis window extension was applied to baseline, as described in the SAP. If a subject received any rescue therapy, the data at/after receipt of rescue therapy are considered as non-responders. Subjects with missing results are considered as non-responders.
Time Frame: Baseline, Week 4
Population: ITT population consisted of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 183 | 91
Participants | 68 | 9
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures were reported and continued when previous outcome measure was statistically significant at two-sided 0.05; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 27.9, 95% CI 2-sided [18.4 to 37.5] — Strata adjusted percentage difference was obtained using weighted average of stratum-specific percentage using CMH

7. Secondary Outcome: Number of Participants With PP NRS < 2 at Week 4
Description: The Peak Pruritus NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores were provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome. Weekly values are calculated as average of 7 consecutive days data up to the target study day (excluding) and set to missing, if less than 4 days data are available. If a subject received any rescue therapy, the data at/after receipt of rescue therapy are considered as non-responders. Subjects with missing results are considered as non-responders.
Time Frame: Week 4
Population: ITT population consisted all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 183 | 91
Participants | 36 | 2
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata-adjusted percentage difference = 18.8, 95% CI 2-sided [12.0 to 25.7] — Strata adjusted percentage difference was obtained using weighted average of stratum-specific percentage using CMH

8. Secondary Outcome: Number of Participants With Adverse Events, Treatment Emergent Adverse Events (TEAEs), Adverse Events of Special Interest (AESIs), and Serious Adverse Events (SAEs)
Description: AE defined as any untoward medical occurrence in clinical study participant administered a medicinal product which does not necessarily have causal relationship with this treatment. TEAEs defined as AEs occurring after first administration of study drug until the last study visit. SAE was any untoward medical occurrence, in view of either Investigator or Sponsor, that resulted in death, was life-threatening, resulted in inpatient hospitalisation or prolongation of existing hospitalisation, resulted in persistent or significant disability/incapacity, was congenital anomaly/birth defect or was important medical event. AESI was noteworthy TEAE for study drug that was to be monitored closely and reported promptly. Relatedness to study drug was based on Investigator's discretion. Analysis was performed on safety population which included all randomised participants who received at least 1 administration of study drug.
Time Frame: From baseline up to end of treatment period (16 Weeks)
Population: Safety population included all randomized participants who received at least 1 administration of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 183 | 91
Participants
  Treatment Emergent Adverse Events (TEAEs) | 112 | 48
  Adverse Events of Special Interest (AESIs) | 21 | 9
  Serious Adverse Events (SAEs) | 4 | 5

ADVERSE EVENTS:
Time Frame: From baseline up to end of treatment period (16 Weeks)
Description: Safety population included all randomized participants who received at least 1 administration of study drug. TEAEs during Treatment period are defined as adverse events with onset date on or after the first dose date till 4 weeks after the last treatment or early discontinuation date whichever is earlier.
Arm/Group | Nemolizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/91
Serious Adverse Events (participants affected / at risk) | 4/183 | 5/91
Other Adverse Events (participants affected / at risk) | 29/183 | 13/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemolizumab (N=183) | Placebo (N=91)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemolizumab (N=183) | Placebo (N=91)
Headache (Nervous system disorders) | 12 (17) | 4 (4)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 10 (15) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 7 (7) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT04501679/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT04501679/SAP_001.pdf